CLINICAL TRIAL: NCT00806442
Title: Treatment of Bronchial Asthma With Borage and Echium Seed Oils
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Wake Forest University Health Sciences (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elliot Israel, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008p001696; P50AT002782 (NIH)
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2017-07-03 (Actual); Last update posted 2017-07-03 (Actual); Status verified 2017-06

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Fatty acids; Leukotrienes; Diet
MeSH Terms: conditions — Asthma | interventions — borage oil; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Borage Seed Oil and Echium Seed Oil (Experimental): Borage/Echium plant seed oils: 2 g/day of borage seed oil and 7 g/day of echium seed oil to provide 1.6 g/day of GLA and 0.9 g/day of SDA.
  Interventions: Drug: Borage Seed Oil and Echium Seed Oil
- 2: Placebo Comparator (Placebo Comparator): Placebo comparator: 9 g/day corn oil
  Interventions: Dietary Supplement: Corn Oil

INTERVENTIONS:
Drug: Borage Seed Oil and Echium Seed Oil — 2 g/day of borage seed oil and 7 g/day of echium seed oil to provide 1.6 g/day of GLA and 0.9 g/day of SDA.
  Other Names: CROSSENTIAL GLA TG40; INCROMEGA V3
  Arms: 1: Borage Seed Oil and Echium Seed Oil
Dietary Supplement: Corn Oil — 9 g/day of corn oil
  Arms: 2: Placebo Comparator

SUMMARY:
The aim of this trial is to determine the efficacy of a combination of two botanicals oils, borage seed oil and echium seed oil, as a potential treatment for bronchial asthma.

DETAILED DESCRIPTION:
Leukotrienes are important in the pathogenesis of inflammation, and leukotriene modifying drugs are now an established treatment for bronchial asthma and rhinitis. Drugs that inhibit the biosynthesis of leukotrienes are likely to be more effective than the currently available drugs that antagonize a single leukotriene receptor. Dietary supplementation with gamma linolenic acid (GLA) in borage seed oil provides effective inhibition of leukotriene generation but also increases circulating free arachidonic acid (AA), which has pro-inflammatory potential. The n-3 fatty acid, eicosapentaenoic acid (EPA), prevented the conversion of GLA to AA. However, EPA is extracted from fish oil, is not well-tolerated due to its taste, and at higher doses appeared to blunt the inhibition of leukotriene biosynthesis by GLA. Stearidonic acid (SDA) is a precursor of EPA that is extracted from Echium plantagineum; it is converted to EPA in humans and it does not have the organoleptic properties of EPA.

We recently completed a dose-ranging study in which we determined the dose of SDA that is sufficient to inhibit the rise in circulating levels of arachidonic acid while maintaining effective inhibition of leukotriene generation.

The goal of the present study is to test the efficacy of dietary supplementation with GLA and SDA (provided in borage seed oil and echium seed oil) in treating bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchial asthma
* Male or female 18 years to 65 years of age
* FEV1 50 to 90% of predicted, or personal best.
* Improvement of >=12% FEV1 with bronchodilator

Exclusion Criteria:

* Pregnant or nursing
* Smoking history of > 10 pack years or active smoking within the past year.
* Due to possible effects on leukotriene biosynthesis, use of the following asthma treatments within the preceding month will be exclusion criteria:

  * leukotriene modifying drugs,
  * theophylline
  * oral steroids.
  * dietary supplements with fatty acids or other products that may interfere with leukotriene generation.
* Treatment within the previous three months with omalizumab (monoclonal antibody directed against IgE)
* Subjects will not be permitted to take non-steroidal anti-inflammatory drugs in the week prior to any measurements of ex vivo leukotriene generation because of their effects on leukotriene biosynthesis via inhibition of prostaglandin generation.
* A history of aspirin-sensitive asthma
* Significant abnormalities in CBC, differential white cell count, renal function, and liver function, or urinalysis.
* Any serious co-morbid medical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Asthma Research Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] James MJ, Ursin VM, Cleland LG. Metabolism of stearidonic acid in human subjects: comparison with the metabolism of other n-3 fatty acids. Am J Clin Nutr. 2003 May;77(5):1140-5. doi: 10.1093/ajcn/77.5.1140. PMID 12716664
- [Background] Chilton-Lopez, Surette ME, Swan DD, Fonteh AN, Johnson MM, Chilton FH. Metabolism of gammalinolenic acid in human neutrophils. J Immunol. 1996 Apr 15;156(8):2941-7. PMID 8609415
- [Background] Johnson MM, Swan DD, Surette ME, Stegner J, Chilton T, Fonteh AN, Chilton FH. Dietary supplementation with gamma-linolenic acid alters fatty acid content and eicosanoid production in healthy humans. J Nutr. 1997 Aug;127(8):1435-44. doi: 10.1093/jn/127.8.1435. PMID 9237935
- [Background] Barham JB, Edens MB, Fonteh AN, Johnson MM, Easter L, Chilton FH. Addition of eicosapentaenoic acid to gamma-linolenic acid-supplemented diets prevents serum arachidonic acid accumulation in humans. J Nutr. 2000 Aug;130(8):1925-31. doi: 10.1093/jn/130.8.1925. PMID 10917903
- [Background] Surette ME, Koumenis IL, Edens MB, Tramposch KM, Chilton FH. Inhibition of leukotriene synthesis, pharmacokinetics, and tolerability of a novel dietary fatty acid formulation in healthy adult subjects. Clin Ther. 2003 Mar;25(3):948-71. doi: 10.1016/s0149-2918(03)80116-9. PMID 12852710
- [Background] Surette ME, Koumenis IL, Edens MB, Tramposch KM, Clayton B, Bowton D, Chilton FH. Inhibition of leukotriene biosynthesis by a novel dietary fatty acid formulation in patients with atopic asthma: a randomized, placebo-controlled, parallel-group, prospective trial. Clin Ther. 2003 Mar;25(3):972-9. doi: 10.1016/s0149-2918(03)80117-0. PMID 12852711
- [Derived] Kazani S, Arm JP, Boyce J, Chhay H, Dutile S, Wechsler ME, Govindarajulu U, Ivester P, Ainsworth HC, Sergeant S, Chilton FH, Israel E. LTC4 synthase polymorphism modifies efficacy of botanical seed oil combination in asthma. Springerplus. 2014 Nov 6;3:661. doi: 10.1186/2193-1801-3-661. eCollection 2014. PMID 25485197
- See also: Asthma Research Center, Brigham and Women's Hospital — http://asthmabwh.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 subjects were enrolled and signed consent; however, only 39 were randomized into a treatment group. 3 subjects screen failed and 1 subject was lost to follow up prior to randomization.
Groups:
- 1 - Borage Seed Oil and Echium Seed Oil, Then Placebo: Borage/Echium plant seed oils: 6.0 g/day borage seed oil and 6.0 g/day echium seed oil) (containing totals of ~ 1.7 g/day of GLA and 0.7 g/day of SDA) 3x day for 3 weeks followed a 3-week washout period, then Placebo (11 g/day corn oil) 3x day for 3 weeks.
- 2 - Placebo, Then Borage Seed Oil and Echium Seed Oil: Placebo (11 g of corn oil/day) 3x day for 3 weeks followed by a 3-week washout period, then Borage/Echium plant seed oils: 6.0 g/day borage seed oil and 6.0 g/day echium seed oil) (containing totals of ~ 1.7 g/day of GLA and 0.7 g/day of SDA) 3x day for 3 weeks.
Period: Overall Study
Arm/Group | 1 - Borage Seed Oil and Echium Seed Oil, Then Placebo | 2 - Placebo, Then Borage Seed Oil and Echium Seed Oil
Started | 18 | 21
First Intervention (3 Wks) | 18 | 21
Washout (3 Wks) | 15 | 14
Second Intervention (3 Wks) | 15 | 14
Completed | 14 | 14
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- All Study Particpants: Includes patients scheduled to receive Borage and Echium seed oil first and participants scheduled to receive placebo first.
Arm/Group | All Study Particpants
Number analyzed (Participants) | 39
Age, Customized [Median (Full Range); unit: years]
  Age | 43 [22 to 64]
Age, Customized [Count of Participants; unit: Participants]
  Age Category: <=18 years | 0
  Age Category: Between 18 and 65 years | 39
  Age Category: >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 27
  Gender: Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced expiratory volume in 1 second (FEV1) in plant seed oil vs. placebo
Time Frame: 6 weeks
Population: Includes participants that completed the study.
Measure: Mean (95% Confidence Interval); unit: liters
Groups:
- Plant Seed Oil: Borage/Echium plant seed oils: 6.0 g/day borage seed oil and 6.0 g/day echium seed oil) (containing totals of ~ 1.7 g/day of GLA and 0.7 g/day of SDA)
- Placebo: Placebo (11 g of corn oil/day)
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 28 | 28
liters | 2.31 [2.22 to 2.39] | 2.25 [2.17 to 2.34]

2. Secondary Outcome: Positive FEV1 Percent Predicted Change Among C Allele Carriers and A Homozygotes
Description: Number of participants with positive change in FEV1 % predicted (>0%) among C allele carriers and A homozygotes in each arm
Time Frame: 6 weeks on each treatment assignment
Population: Patients who are C allele carriers or A homozygotes
Measure: Count of Participants; unit: Participants
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  C-allele Carriers: number analyzed (Participants) | 9 | 9
  C-allele Carriers | 6 | 2
  A Homozygotes: number analyzed (Participants) | 19 | 19
  A Homozygotes | 11 | 10

3. Secondary Outcome: Peak Flow Rate (PEFR)
Description: Morning Peak Flow Rate in plant seed oil vs. placebo
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: liters/minute
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 28 | 28
liters/minute | 337.13 [328.43 to 345.82] | 339.34 [330.65 to 348.04]

4. Secondary Outcome: Frequency of Rescue Use of Short Acting Beta-2 Agonists
Description: Average number of puffs of albuterol daily in plant seed oil vs. placebo
Time Frame: 6 weeks
Population: one participant is missing some data on this measure
Measure: Mean (95% Confidence Interval); unit: Avg number of puffs of albuterol daily
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 27 | 27
Avg number of puffs of albuterol daily | 0.69 [0.42 to 0.97] | 0.50 [0.23 to 0.78]

5. Secondary Outcome: Day-time Symptoms of Bronchial Asthma
Description: Day-time symptom scores in plant seed oil vs. placebo. 0 = Absent: No symptoms
  1. = Mild: Symptom did not interfere with normal daily activity or sleep
  2. = Moderate: Symptom was sufficient to interfere with normal daily activity or sleep
  3. = Severe: Symptom was so severe as to prevent normal daily activity or sleep
  These numbers were used for 1. Shortness of breath 2. Chest tightness 3. Wheezing 4. Cough 5. Phlegm/Mucus.
  The total score is the sum of the 5 item scores, for a range of 0-15. A higher score represents more severe symptoms. Each participant's score is the average of varying numbers of diary cards. The treatment phase visits at 6 weeks consisted of 3 weeks of diary cards with a +/- 5 day window. The baseline visits had 2 weeks of diary cards with a +/- 5 day window. The treatment phase measures are adjusted for the baseline measures.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | 2.51 [1.79 to 3.22] | 1.61 [0.90 to 2.33]

6. Secondary Outcome: Night-time Wakenings
Description: Average number of night-time wakenings in plant seed oil vs. placebo
Time Frame: 6 weeks
Population: one participant is missing some night-time wakening data
Measure: Mean (95% Confidence Interval); unit: average number of night-time wakenings
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 27 | 27
average number of night-time wakenings | 0.16 [0.05 to 0.27] | 0.13 [0.02 to 0.23]

7. Secondary Outcome: Urinary Leukotriene Levels
Description: Urinary leukotriene levels in plant seed oil vs. placebo
Time Frame: 6 weeks
Population: one participant was missing some urinary leukotriene data
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Plant Seed Oil | Placebo
Number analyzed (Participants) | 27 | 27
ng/ml | 0.101 [0.085 to 0.117] | 0.088 [0.072 to 0.105]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for one year.
Description: Adverse events data were collected for one year, from the time of first patient enrollment to the last date of adverse event resolution.
Groups:
- Washout After Plant Seed Oil: Washout period between first (plant seed oil) and second (placebo) treatment assignments
- Washout After Placebo: Washout period between first (placebo) and second (plant seed oil) treatment assignments
Arm/Group | Plant Seed Oil | Placebo | Washout After Plant Seed Oil | Washout After Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 13/28 | 14/28 | 6/14 | 5/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plant Seed Oil (N=28) | Placebo (N=28) | Washout After Plant Seed Oil (N=14) | Washout After Placebo (N=14)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — subject experienced phlegm, cough, and wheeze during washout phase
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plant Seed Oil (N=28) | Placebo (N=28) | Washout After Plant Seed Oil (N=14) | Washout After Placebo (N=14)
Drop in Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
drop in hematocrit (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
stomach ache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urticaria (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
uterine fibroid (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7) | 4 (5) | 2 (2)
cough, chest tightness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
worsening asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
bruised rib (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No